CLINICAL TRIAL: NCT00536341
Title: A Phase I/II Study of Fludarabine, Rituximab, and Lenalidomide in Minimally Treated and Untreated Patients With Chronic Lymphocytic Leukemia
Brief Title: Fludarabine, Rituximab, and Lenalidomide in Minimally Treated/Untreated Patients With Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Celgene Corporation (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI CLL 02
Record Dates: First submitted 2007-09-24; First posted 2007-09-27 (Estimated); Results first posted 2016-05-04 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; untreated; minimally treated; fludarabine; rituximab; lenalidomide
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Lenalidomide; Rituximab; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- lenalidomide, fludarabine, rituximab (Experimental): Phase I Non-stratified, dose-escalation: >=3 patients per dose level. Safety and tolerability will be evaluated every 2 weeks during the active treatment. Doses of lenalidomide will be escalated, while the fludarabine and rituximab doses remain fixed.
  Phase II The Phase II regimen will be chosen following a review of the Phase I data. Following selection of the Phase II schedule, 40 treatment naive patients will be enrolled and treated with the Phase II regimen every 28 days for up to 6 courses. For those patients achieving a CR after 3 cycles, one additional cycle of treatment will be administered beyond CR confirmation.
  Interventions: Drug: lenalidomide; Drug: Rituximab; Drug: Fludarabine

INTERVENTIONS:
Drug: lenalidomide — 2.5 mg orally (PO) daily, Days 8-28, Cycle 1; 5.0 mg PO daily, Days 8-28 Cycles 2-6
  Other Names: Revlimid
Drug: Rituximab — 375 mg/m2 Cycle 1 (split over Day 1 & Day 2); 500 mg/m2 Day 1 of Cycles 2-6
  Other Names: Rituxan
Drug: Fludarabine — 25 mg/m2 on Days 1, 2, and 3
  Other Names: Fludara

SUMMARY:
This phase I/II trial will combine fludarabine, rituximab, and lenalidomide in untreated or minimally treated (Phase I only) CLL patients, employing fixed doses of fludarabine and rituximab, using a schedule similar to that examined by investigators at MD Anderson (J Clin Oncol 23(18):4079-88, 2005). Given that the optimal dose and schedule is not currently known, this trial will perform a phase I component followed by a phase II examination to further explore this regimen's activity.

DETAILED DESCRIPTION:
While progress has been made in treating CLL patients over the last decade, a cure remains elusive for many patients treated with standard therapies. The combination of fludarabine, a purine analog, and rituximab, a monoclonal antibody, is an effective and frequently used therapy for CLL. However, this drug combination is associated with increased toxicity. Lenalidomide has been shown to be less toxic and has been used to treat hematologic malignancies including CLL. We propose this Phase I/Phase II study to examine the combination of lenalidomide with a rituximab/fludarabine backbone.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Age >=18 years at the time of signing the informed consent form.
* Patient must have histopathologically confirmed B-cell CLL
* For Phase I only: Untreated or minimally treated patients (patients who have received only prior single agent rituximab) are eligible. For those patients who have had rituximab monotherapy, last dose must be greater than 90 days prior to beginning study treatment.
* For Phase II only: Untreated B-cell CLL patients only.
* Rai staging, will be employed. Patients must have Rai stage III/IV disease (irrespective of symptoms) OR symptomatic Rai stage 0-II disease, requiring therapy as defined by NCI 1996 guidelines.
* Platelets must be > 75,000/mm3 and absolute neutrophil count must be > 1000/mm3 within 14 days of starting protocol treatment unless treating physicians deems the neutropenia is related to marrow involvement and then ANC > 750/mm3 is allowed.
* Serum creatinine <=2.0 mg/dl obtained within 14 days of starting protocol treatment. Creatinine clearance as determined by the Cockroft-Gault formula, using ideal body weight, must be > 30 mL/minute.
* AST or ALT must be < 3 x the upper limit of normal within 14 days of starting treatment.
* ECOG performance of 0, 1 or 2.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL within 10 - 14 days prior to and again within 24 hours of starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* Disease free of prior malignancies for >= 2 years (including carcinoma in situ of the cervix or breast) treated with curative intent and anticipated 5 year disease-free survival is greater than 90%. Any basal cell or squamous cell carcinoma of the skin treated with curative intent is permitted.
* Able to take aspirin (325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use low molecular weight heparin).

Exclusion Criteria:

* Major surgery less than 28 days prior to study treatment.
* Any prior use of lenalidomide or thalidomide.
* Concurrent use of other anti-cancer therapies.
* Pregnant or breast feeding females. (Lactating females may be considered if they agree not to breast feed while receiving study treatment and until 12 months following last dose of rituximab).
* History of pulmonary embolus or deep vein thrombosis.
* Clinically significant heart dysfunction, defined as New York Heart Association class III or IV, at the time of screening, or history of myocardial infarction or heart failure within 6 months preceding the first study treatment (cardiac ejection fraction must be >= 50% within 8 weeks of beginning study treatment for any patient with a history of clinically significant heart dysfunction).
* Known positive for HIV, hepatitis B surface Ag, hepatitis B core antibody, or hepatitis C. Mandatory testing is not required, but should be considered in patients deemed high risk or suspicious.
* Active infection requiring oral or intravenous antibiotics at study entry. After infection resolves patient may be evaluated for enrollment.
* Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenia purpura.
* Richter's transformation.
* CNS involvement.
* Other severe, acute, or chronic medical or psychiatric condition, laboratory abnormality, or difficulty complying with protocol requirements that may increase the risk associated with study participation or study drug administration or may interfere with interpretation of study results that in the judgment of the investigator would make the patient inappropriate for this study or that would prevent the patient from signing the informed consent form.
* Use of any other biologic agent or disease-modifying anti-rheumatic drugs (DMARDS).
* Known anaphylaxis or IgE-mediated hypersensitivity to murine proteins or any component of rituximab.
* Evidence of laboratory TLS by Cairo-Bishop criteria (subjects may be enrolled upon correction of electrolyte abnormalities).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-01; Primary Completion 2013-04 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian W. Flinn, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (6):
- United States (6):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - South Carolina Oncology Associates, PA, Columbia, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee

REFERENCES:
- See also: Sarah Cannon Research Institute — http://www.sarahcannonresearch.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Level 1: Rituximab 375 mg/m^2 cycle 1 (split over Day 1 & Day 2), 500 mg/m^2 Day 1 of cycles 2-6 Fludarabine 25 mg/m^2 on days 1, 2 and 3 Lenalidomide 2.5 mg PO daily Days 8-28 all cycles 1-6
- Dose Level 2: Rituximab 375 mg/m^2 cycle 1 (split over Day 1 & Day 2), 500 mg/m^2 Day 1 of cycles 2-6 Fludarabine 25 mg/m^2 on days 1, 2 and 3 Lenalidomide 2.5 mg PO daily Days 8-28 cycle 1, 5.0 mg PO days 8-28 cycles 2-6
Period: Overall Study
Arm/Group | Dose Level 1 | Dose Level 2
Started | 10 | 54
Completed | 5 | 43
Not Completed | 5 | 11

BASELINE CHARACTERISTICS:
Population: All enrolled and treated patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1 | Dose Level 2 | Total
Number analyzed (Participants) | 10 | 54 | 64
Age, Continuous [Median (Full Range); unit: years] | 67 [49 to 74] | 63 [44 to 82] | 64 [44 to 82]
Gender [Count of Participants; unit: Participants]
  Female | 2 | 25 | 27
  Male | 8 | 29 | 37
Region of Enrollment [Number; unit: participants]
  United States | 10 | 54 | 64

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events as a Measure of Safety and Tolerability
Description: Recorded from first treatment until 30 days after last treatment and assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: 63 months
Population: All treated patients
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 10 | 54
participants
  Fatigue | 8 | 40
  Neutropenia | 7 | 41
  Anemia | 8 | 34
  Leukopenia | 7 | 34
  Thrombocytopenia | 8 | 30
  Rash | 6 | 27
  Nausea | 7 | 25
  Constipation | 3 | 15
  Anorexia | 4 | 12
  Fever | 3 | 13
  Hyperhidrosis | 3 | 13
  Arthralgia | 1 | 14
  Edema Limbs | 3 | 12
  Pruritus | 0 | 15
  Back pain | 3 | 11
  Headache | 1 | 13
  Chills | 2 | 11
  Insomnia | 2 | 11
  Vomiting | 2 | 11
  Dysgeusia | 1 | 11
  Abdominal Pain | 2 | 9
  Allergic Reaction | 4 | 7
  Diarrhea | 3 | 8
  Cough | 2 | 8
  Dizziness | 2 | 8
  Dyspnea | 0 | 10
  Hypotension | 1 | 9
  Myalgia | 2 | 8

2. Primary Outcome: Complete Response Rate
Description: An improvement in complete response to at least 60% following treatment, assessed using CT scans, clinical/lab examinations, and bone marrow aspirations, as defined by National Cancer Institute Working Group Response Criteria.
Time Frame: At 12 weeks during treatment and 2 months post-treatment until disease progression, projected 8 months
Population: All patients deemed evaluable and evaluated for response
Measure: Number; unit: participants
Arm/Group | Dose Level 1 | Dose Level 2
Number analyzed (Participants) | 9 | 41
participants | 4 | 9

3. Secondary Outcome: Progression-Free Survival
Description: Measured from first treatment to disease progression and assessed using Kaplan-Meier methods.
Time Frame: Every 3 months during treatment until disease progression and every 6 months thereafter, up to 5 years
Population: All treated patients, all dose levels
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients
Number analyzed (Participants) | 64
months | 24.64 [21.125 to NA] — Not reached at this time

4. Secondary Outcome: Overall Survival
Description: Defined as the time from Day 1 of treatment administration to date of death from any cause, estimated using Kaplan-Meier methods.
Time Frame: Every 3 months until treatment discontinuation, expected average of 6 months and then every 6 months thereafter up to 5 years
Population: All treated patients, all dose levels
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | All Patients
Number analyzed (Participants) | 64
months | NA [NA to NA] — Median OS not reached at this time

ADVERSE EVENTS:
Time Frame: 63 months
Arm/Group | Dose Level 1 | Dose Level 2
Serious Adverse Events (participants affected / at risk) | 2/10 | 16/54
Other Adverse Events (participants affected / at risk) | 10/10 | 54/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=10) | Dose Level 2 (N=54)
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Allergic Reaction (Immune system disorders) | 0 | 1
Bronchial Infection (Infections and infestations) | 0 | 2
Chills (General disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Edema limbs (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Fever (General disorders) | 0 | 2
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Infections and infestations - Other, gastrointestinal infection NOS (Infections and infestations) | 0 | 1
Infections and infestations - Other, pneumonia (Infections and infestations) | 1 | 1
Infections and infestations - Other, unspecified (Infections and infestations) | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1
Mucositis (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Sepsis (Infections and infestations) | 0 | 1
Tumor Lysis Syndrome (Metabolism and nutrition disorders) | 0 | 1
White blood cell decreased (Investigations) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=10) | Dose Level 2 (N=54)
Fatigue (General disorders) | 8 | 40
Neutrophil count decreased (Investigations) | 7 | 41
Anemia (Blood and lymphatic system disorders) | 8 | 34
White blood cell decreased (Investigations) | 7 | 34
Platelet count decreased (Investigations) | 8 | 30
Rash (Skin and subcutaneous tissue disorders) | 6 | 27
Nausea (Gastrointestinal disorders) | 7 | 25
Constipation (Gastrointestinal disorders) | 3 | 15
Anorexia (Metabolism and nutrition disorders) | 4 | 12
Fever (General disorders) | 3 | 13
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 14
Edema limbs (General disorders) | 3 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 11
Headache (Nervous system disorders) | 1 | 13
Chills (General disorders) | 2 | 11
Insomnia (Psychiatric disorders) | 2 | 11
Vomiting (Gastrointestinal disorders) | 2 | 11
dysgeusia (Nervous system disorders) | 1 | 11
Abdominal pain (Gastrointestinal disorders) | 2 | 9
Allergic reaction (Immune system disorders) | 4 | 7
Diarrhea (Gastrointestinal disorders) | 3 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Dizziness (Nervous system disorders) | 2 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 10
Hypotension (Vascular disorders) | 1 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 7
Aspartate aminotransferase increased (Investigations) | 0 | 8
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 7
Hyperkalemia (Metabolism and nutrition disorders) | 2 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 7
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Sinusitis (Infections and infestations) | 0 | 7
Alanine aminotransferase increased (Investigations) | 1 | 5
Alkaline phosphatase increased (Investigations) | 1 | 5
Mucositis (Gastrointestinal disorders) | 0 | 6
Dehydration (Metabolism and nutrition disorders) | 0 | 5
depression (Psychiatric disorders) | 0 | 5
Infections and infestations - Other, unspecified (Infections and infestations) | 1 | 4
Investigations - Other, LDH increased (Investigations) | 0 | 5
Tremor (Nervous system disorders) | 1 | 4
Blood bilirubin increased (Investigations) | 0 | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 4
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 4
Hyponatremia (Metabolism and nutrition disorders) | 1 | 3
Skin and subcutaneous tissue disorders - Other, erythema (Skin and subcutaneous tissue disorders) | 3 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Upper respiratory infection (Infections and infestations) | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites